CLINICAL TRIAL: NCT04188561
Title: Comparative Study Between Intra Articular Injection of Hyaluronic Acid (HA) With Platelet Rich Plasma (PRP) Versus Genicular Nerve Thermal Radiation in Management of Pain in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32094/01/18
Record Dates: First submitted 2019-11-17; First posted 2019-12-06 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This Prospective randomized study was conducted on (100) knees with mild to moderate osteoarthritis and scheduled for Intra articular injection or Genicular nerve radiofrequency at Tanta University Hospital (Intra articular injection was done in pain clinic and Radiofrequency was done in operating room
Who Masked: Participant, Care Provider
Masking Description: Closed Opauqe Envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraarticular injection Group (Active Comparator): Patients included in the study had been received 2 ml hyaluronic acid with concentration of 22mg/ml . Platelet rich plasma is arranged by withdrawing 10 ml of patient's personal venous blood, anticoagulant is added, and centrifuged by duo-spin method, at the rate of 3500 rpm for five minutes then injected twice with 2 weeks interval
  Interventions: Drug: Intra articular injection Group
- Radiofrequency Group (Active Comparator): Radiofrequency Generator is a four electrode pain management for interventional pain management procedures. Patients had been placed in the supine position and their knee will be supported by a small pillow placed beneath the popliteal fossa. Fluoroscopic images of knee joint had been obtained. Possible locations of genicular nerves had been determined on the lateral, medial aspects of the lower end of the femoral bone and on the medial aspect of the tibia, under fluoroscopic guidance.
  Interventions: Device: Radiofrequency Group

INTERVENTIONS:
Drug: Intra articular injection Group — Patients included in the study had been received 2 ml high molecular weight (1.476 x 106 average Daltons) hyaluronic acid with concentration of 22mg/ml (OPTIVISC UK hyaluronic acid for intra articular injection). Platelet rich plasma is arranged by withdrawing 10 ml of patient's personal venous blood, anticoagulant is added, and centrifuged by duo-spin method, at the rate of 3500 rpm for five minutes then injected twice with 2 weeks interval. 3 distinct layers are produced by the end of the centrifugation: plasma, buffy coat (platelet) and RBCs, about 3 - 3.5 ml of PRP is produced
  at the end with platelet concentration of 1.4 - 1.6 million/μl on average.
  Other Names: Intra articular injection of hyaluronic acid and platelet rich plasma
  Arms: Intraarticular injection Group
Device: Radiofrequency Group — Thermal radiation is done by Neurotherm 2000 (Neurotherm NT 2000 Radiofrequency (RF) Generator is a four electrode pain management (RF) generator for interventional pain management procedures. Neurotherm's newest system offers accurate independent controls of each electrode through the touch screen interface and output control knobs.), Patients from the radiofrequency (RF) group had been placed in the supine position and their knee will be supported by a small pillow placed beneath the popliteal fossa. Fluoroscopic images of knee joint had been obtained. Possible locations of genicular nerves had been determined on the lateral, medial aspects of the lower end of the femoral bone and on the medial aspect of the tibia, under fluoroscopic guidance.
  Other Names: Thermal radiation of Genicular nerve
  Arms: Radiofrequency Group

SUMMARY:
Intraarticular injection (IAI) of Platelet rich plasma (PRP) with Hyaluronic acid (HA) Versus Radiofrequency (RF) of genicular nerve for pain reduction of of knee osteoarthritis , Improving daily activity and reduction analgesia requirements

DETAILED DESCRIPTION:
In this study the investigators to comparing between the effect of Intra articular injection of hyaluronic acid (HA) with platelet rich plasma (PRP) versus genicular nerve thermal radiation in management of pain in knee osteoarthritis.

Knee assessment and pain score recorded according to Visual Analogue Scale (VAS) after one week, one month, three months, six months following intraarticular injection and radiation.

All analgesics stopped and only (Arcoxia "etoricoxib" 60 mg, 90 mg) was taken after the procedure, total day dose and frequency will be reported, other analgesics taken by the patient is reported also.

Improvement of daily activities and clinical examination for the studied knees is observed.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Knee osteoarthritis.
* Body mass index: 24 - 42 kg/m2

Exclusion Criteria:

* Coagulopathy.
* Acute local or systemic infections with knee effusion Previous knee surgery (relative Contraindication).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Pain Measurment via Visual analogue score | Measured throuout 6 months follow up session
  Visual analogue score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity was measured throuout 6 months follow up session

SECONDARY OUTCOMES:
Analgesic requirements Comparison | Throuout 6 months follow up session
  Compairing between analgesia requirements in Rf group and IAI group
Improvement of daily activities between 2 groups | Throuout 6 months follow up session
  Compairing between analgesia requirements in Rf group and IAI group

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Publication